CLINICAL TRIAL: NCT02722915
Title: Symptom Based Treatment Affects Brain Plasticity - the Role of Verbal Auditory Hallucinations
Acronym: APIC-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-139
Record Dates: First submitted 2016-03-10; First posted 2016-03-30 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2019-09

CONDITIONS: Hallucinations, Verbal Auditory
Keywords: fMRI; neurofeedback; hallucination; schizophrenia
MeSH Terms: conditions — Hallucinations; Schizophrenia | interventions — Neurofeedback; Gene Expression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fMRI Neurofeedback up-regulation (Experimental): Study related procedures included: PANAS, AVHRS, SF 36 (questionnaires or evaluations)
  Interventions: Procedure: fMRI; Behavioral: Neurofeedback; Other: PANAS; Other: AVHRS; Other: SF36
- fMRI Neurofeedback down-regulation (Experimental): Study related procedures included: PANAS, AVHRS, SF 36 (questionnaires or evaluations)
  Interventions: Procedure: fMRI; Behavioral: Neurofeedback; Other: PANAS; Other: AVHRS; Other: SF36

INTERVENTIONS:
Procedure: fMRI — collection of functional brain data for 1 hour per day
  Other Names: functional magnetic resonance imaging
Behavioral: Neurofeedback — Task of the participants is to increase or decrease the connectivity between selected brain regions in double-blind, randomized order. After the regulation they will get a feedback about the regulation success. (Patients and controls with AVH: days 3 & 4; controls without AVH: Days 2 & 3)
Other: PANAS — to assess the mood before and after the fMRI and after 1 week during a telephone interview
  Other Names: Positive And Negative Affect Scales
Other: AVHRS — to assess the intensity and quality of the hallucinations before and after the fMRI and after 1 week during a telephone interview
  Other Names: Auditory Vocal Hallucinations Rating Scale
Other: SF36 — questionnaire about life quality after 1 week during a telephone interview

SUMMARY:
The aim of the study is the examination of brain plasticity on verbal auditory hallucinations (AVH) after neuromodulation with fMRI (functional magnetic resonance imaging) neurofeedback. During the training of fMRI neurofeedback subjects are trained to regulate consciously the connectivity of areas which are associated with hallucinations.The aim is to improve perceived hallucinations' intensity in everyday life of the patients as well as investigating the impact of neurofeedback on resting-state networks in the brain. As control groups, control subjects without AVH and participants with AVH, but no psychiatric diagnosis will be included.

DETAILED DESCRIPTION:
This study investigates the brain plasticity after neuromodulation with fMRI neurofeedback on verbal auditory hallucinations (AVH). The new technique of real-time fMRI enables subjects to influence their brain activity in certain areas based on neurofeedback. Current brain activity as measured by fMRI will be reported to the participants in real time via brain computer interface (BCI). Due to the identification of contingency between feedback and mental strategies subjects are able to control their own brain activity consciously. This provides the opportunity to control symptoms such as AVH. Neurofeedback has been tested on subjects with schizophrenia, leading to conscious control of circumscribed brain areas. Recent studies show that, in addition to the modulation of single areas, neurofeedback can also modulate connectivity between different areas. Thus, it is possible to regulate not only single brain regions but also whole networks.

AVH are a key symptom of schizophrenia. They limit social functions significantly and are resistant to the therapy with antipsychotics in 25 % of cases. AVH also occur in 6-15 % of the healthy population, without meeting any diagnostic criteria for schizophrenia or other psychiatric disorders. This study will perform a direct, not-invasive and selective modulation of networks underlying AVH and assess their neural, cognitive and emotional effects. The focus of this study is on the connectivity between auditory cortex and inferior frontal cortex. Various studies demonstrated that the auditory cortex exhibits an abnormal function in schizophrenia patients. It was shown that during AVH, auditory cortex (superior temporal lobe) and inferior frontal cortex synchronize spontaneously. These regions play an essential role in speech perception and processing. An increased synchronisation of these areas could lead to the development of AVH. This study will try to reduce frontotemporal connectivity to uncouple the regions. Increasing connectivity of both areas will serve as control condition and furthermore intensify the perceived control of the own brain activity and of the associated AVH. Thus, patients will learn which factors influence the appearance of their hallucinations.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia according to ICD-10 (F2x) with verbal hallucinations or only verbal hallucinations (no psychiatric diagnosis) or healthy subjects without verbal hallucinations
* Fluent German language skills

Exclusion Criteria:

* addiction
* severe affective disorder
* any contraindication to MRI examination or claustrophobia
* pregnant or lactating women
* traumatic brain lesions
* acute physical or neurological impairments
* acute suicidal tendency
* Lack of informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
change in self-control over neuronal connectivity | 1 week
  fMRI-BCI as a measure before and after the regulation of the brain activity

SECONDARY OUTCOMES:
Changes from baseline in brain plasticity | 2 weeks
  fMRI as a measure for brain plasticity before and after neurofeedback
Change in pathology (AVH) | 1 week after interventions
  Auditory Vocal Hallucinations Rating Scale (AVHRS) as a measure of the intensity and quality of the hallucinations before and after the fMRI and after 1 week during a telephone interview
number of patients and subjects with benefits from neurofeedback training | 2 weeks
change in brain activation | 1 week after interventions
  fMRI as a measure before and after the following resting state
Change in pathology (mood) | 1 week after interventions
  Positive And Negative Affect Scales (PANAS) as a measure of mood before and after the fMRI and after 1 week during a telephone interview
Change in perceived quality of life | 1 week after interventions
  SF36 questionnaire as a measure of the quality of life before and after the fMRI and after 1 week during a telephone interview

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Mathiak, Prof MD PhD, Principal Investigator — University Hospital RWTH Aachen, Department of Psychiatry, Psychotherapy and Psychosomatics
Locations (1):
- University Hospital RWTH Aachen, Department of Psychiatry, Psychotherapy and Psychosomatics, Aachen, Germany